CLINICAL TRIAL: NCT00852514
Title: The Optimization of Blood Pressure and Fluid Status Control With Eight-Polar Bioelectrical Impedance Analysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Jinn-Yang Chen, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHIRB 95-08-28A
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Hypertension; Fluid Overload; Heart Diseases
Keywords: Bioimpedance; ultrafiltration; blood pressure; pulse pressure
MeSH Terms: conditions — Hypertension; Edema; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Monthly BIA (Experimental): monthly BIA to monitor fluid status
  Interventions: Device: Bioelectrical impedance-guide dry weight reduction

INTERVENTIONS:
Device: Bioelectrical impedance-guide dry weight reduction — for optimal determination of fluid status, monthly BIA was performed to monitor fluid status and avoid dehydration

SUMMARY:
Peritoneal dialysis (PD) is a widely used modality of renal replacement therapy. Due to its continuous nature of therapy, better control of fluid status and preservation of residual renal function were presumed by most nephrologists. However, recent evidences showed that it might not be the case. The severity of fluid overloading and the need for anti-hypertensive agents to control blood pressure seems to be more severe for PD patients. Therefore, more aggressive strategy to control dry weight is mandatory in PD patients. However, over reduction of dry weight might affect residual renal function (RRF) and, probably, the survival of PD patients. A balance between reduction of dry weight and preservation of RRF is crucial for the care of PD patients. Currently, only clinical measures like cardiothoracic ratio on chest X-ray and absence of pedal edema were used to evaluate PD patient's dry weight. There is no objective method to determine dry weight accurately. In this prospective and randomized study, the investigators will use multi-frequency bio-impedance (MF-BIA) to detect intracellular and extracellular water (ECW) content of patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 80

Exclusion Criteria:

* type I DM
* Severe heart failure
* unstable angina

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jinn-Yang Chen, MD, PhD, Principal Investigator — Division of Nephrology, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan